CLINICAL TRIAL: NCT01261975
Title: Co-Axial Micro-incision Cataract Surgery(C-MICS) Versus Standard Co-Axial Small Incision Cataract Surgery Using the Stellaris Enhancement System
Brief Title: Co-Axial Micro-Incision Versus Co-Axial Small Incision Cataract Surgery Using the Stellaris Enhancement System
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 607
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Results first posted 2012-02-27 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-01

CONDITIONS: Cataract; Aphakia
Keywords: Ocular Surgery; Intraocular Lens
MeSH Terms: conditions — Cataract; Aphakia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coaxial Micro-Incision Cataract Surgery (Experimental): 1.8 mm coaxial microincision
  Interventions: Procedure: Coaxial Micro-Incision Cataract Surgery
- Coaxial Small Incision Cataract Surgery (Active Comparator): 2.75 mm standard incision
  Interventions: Procedure: Coaxial Small Incision Cataract Surgery

INTERVENTIONS:
Procedure: Coaxial Micro-Incision Cataract Surgery — 1.8 mm coaxial micro incision
  Other Names: Stellaris Vision Enhancement System
  Arms: Coaxial Micro-Incision Cataract Surgery
Procedure: Coaxial Small Incision Cataract Surgery — 2.75 mm coaxial incision
  Other Names: Stellaris Vision Enhancement System
  Arms: Coaxial Small Incision Cataract Surgery

SUMMARY:
The objective of this study is to test the hypothesis that the time to reach a stable refraction is significantly shorter in eyes operated with the 1.8 mm coaxial microincision compared to eyes operated with the 2.75 mm standard incision using the Stellaris Vision Enhancement System.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be undergoing bilateral primary in-the-bag intraocular lens (IOL) implantation for the correction of aphakia.
* Subject's ocular media must be clear except for the presence of the cataract in both eyes.

Exclusion Criteria:

* Subject with any disease, which, in the Investigator's opinion, might interfere with the conduct of the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Williart, MD, Study Director — Bausch & Lomb Incorporated

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at one clinical site in Europe. First participant was enrolled on 8/25/2009 and last participant exited the study on 4/27/2010. Study lasted six months for enrollment and three months for follow-up.
Pre-assignment Details: 36 participants at least 50 years of age were enrolled in bilateral cataract surgery with phacoemulsification and intraocular lens implantation for the correction of aphakia. The Stellaris Vision Enhancement System was used for a 1.8mm Coaxial Micro-Incision procedure in one eye and a 2.75mm coaxial standard procedure in the contralateral eye.
Groups:
- Cataract Surgery: Cataract surgery with phacoemulsification. Eligible patients were randomized to undergo cataract surgery using the 1.8 mm coaxial micro incision technique in either the right eye or the left eye. The fellow eye was assigned to undergo cataract surgery using the 2.75 mm standard incision. The Stellaris Vision Enhancement System was used for the surgery.
Period: Overall Study
Arm/Group | Cataract Surgery
Started | 36 (36 Participants 72 eyes started)
Completed | 35 (35 Participants 70 eyes completed)
Not Completed | 1
Not completed — Surgical complication | 1

BASELINE CHARACTERISTICS:
Groups:
- Cataract Surgery: Cataract surgery with phacoemulsification using the Stellaris Vision Enhancement System
Arm/Group | Cataract Surgery
Number analyzed (Participants) | 36
Age, Customized [Number; unit: participants]
  Aged 71 to 81 years | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 11
Region of Enrollment [Number; unit: participants]
  Europe | 36

OUTCOME MEASURES:

1. Primary Outcome: Refractive Stability
Description: Cumulative portion of eyes achieving refractive stability within 0.5 D of the final value for the remainder of the trial by surgical procedure and visit.
Time Frame: 12 weeks
Population: Cumulative Proportion of Eyes Achieving Refractive Stability (within 0.5 D)- Full analysis Set (FAS) Population
Measure: Number; unit: Eyes
Units Other Than Participants: eyes
Groups:
- Coaxial Micro-Incision Cataract Surgery: 1.8 mm coaxial micro-incision cataract surgery (C-MICS) with phacoemulsification using the Stellaris Vision Enhancement System
- Coaxial Small-Incision Cataract Surgery: 2.75 mm coaxial standard cataract surgical procedure with phacoemulsification using the Stellaris Vision Enhancement System.
Arm/Group | Coaxial Micro-Incision Cataract Surgery | Coaxial Small-Incision Cataract Surgery
Number analyzed (Participants) | 36 | 35
Number analyzed (eyes) | 36 | 35
Eyes
  Visit 1 | 17 | 23
  Visit 2 | 25 | 25
  Visit 3 | 27 | 27
  Visit 4 | 27 | 28
  Visit 5 | 28 | 30
  Visit 6 | 29 | 31
  Visit 7 | 29 | 33

2. Secondary Outcome: Best Corrected Visual Acuity
Description: Best corrected distance visual acuity(BCVA) was assessed using logMAR charts. Change from preoperative visit summarized by visit. A minus change represents an improvement of the visual acuity
Time Frame: Visit 1, visit 2, visit 3, visit 4
Population: Best Corrected Distance Visual Acuity (logMAR), Change from baseline, FAS Population
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Coaxial Micro-Incision Cataract Surgery | Coaxial Small-Incision Cataract Surgery
Number analyzed (Participants) | 36 | 35
Number analyzed (eyes) | 36 | 35
logMAR
  Visit 1 | -0.26 (0.24) | -0.27 (0.29)
  Visit 2 | -0.37 (0.22) | -0.39 (0.26)
  Visit 3 | -0.38 (0.20) | -0.38 (0.27)
  Visit 4 | -0.39 (0.24) | -0.38 (0.27)

3. Secondary Outcome: Best Corrected Visual Acuity
Description: Best corrected distance visual acuity(BCVA) was assessed using logMAR charts. Change from baseline summarized by visit. A minus change represents an improvement of the visual acuity.
Time Frame: visit 5, visit 6, visit 7, visit 8
Population: Best Corrected Distance Visual Acuity (logMAR), change from baseline, FAS Population
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Coaxial Micro-Incision Cataract Surgery | Coaxial Small-Incision Cataract Surgery
Number analyzed (Participants) | 35 | 35
Number analyzed (eyes) | 35 | 35
logMAR
  Visit 5 | -0.40 (0.22) | -0.40 (0.27)
  Visit 6 | -0.39 (0.24) | -0.42 (0.27)
  Visit 7 | -0.40 (0.24) | -0.42 (0.26)
  Visit 8 | -0.41 (0.22) | -0.41 (0.28)

4. Secondary Outcome: Uncorrected Visual Acuity
Description: Uncorrected visual acuity(UCVA) was assessed using logMAR charts. Change from baseline summarized by visit.
Time Frame: Visit 1, visit 2, visit 3, visit 4
Population: Uncorrected Visual Acuity (logMAR), change from baseline, FAS Population
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Coaxial Micro-Incision Cataract Surgery | Coaxial Small-Incision Cataract Surgery
Number analyzed (Participants) | 36 | 35
Number analyzed (eyes) | 36 | 35
logMAR
  Visit 1 | -0.22 (0.32) | -0.34 (0.31)
  Visit 2 | -0.37 (0.29) | -0.45 (0.31)
  Visit 3 | -0.37 (0.30) | -0.41 (0.32)
  Visit 4 | -0.36 (0.30) | -0.46 (0.31)

5. Secondary Outcome: Uncorrected Visual Acuity
Description: Uncorrected visual acuity(UCVA) was assessed using logMAR charts. Change from baseline summarized by visit.
Time Frame: visit 5, visit 6, visit 7, visit 8
Population: Uncorrected Visual Acuity (logMAR), change from baseline, FAS Population
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Coaxial Micro-Incision Cataract Surgery | Coaxial Small-Incision Cataract Surgery
Number analyzed (Participants) | 35 | 35
Number analyzed (eyes) | 35 | 35
logMAR
  Visit 5 | -0.36 (0.33) | -0.48 (0.32)
  Visit 6 | -0.35 (0.31) | -0.47 (0.34)
  Visit 7 | -0.36 (0.35) | -0.49 (0.33)
  Visit 8 | -0.38 (0.31) | -0.51 (0.32)

6. Secondary Outcome: Surgically Induced Astigmatism (SIA)
Description: Surgically induced astigmatism was presented in dioptres at each visit.
Time Frame: Visits 1-3
Population: Surgically Induced Astigmatism, FAS Population
Measure: Mean (Standard Deviation); unit: Dioptres
Units Other Than Participants: eyes
Arm/Group | Coaxial Micro-Incision Cataract Surgery | Coaxial Small-Incision Cataract Surgery
Number analyzed (Participants) | 36 | 35
Number analyzed (eyes) | 36 | 35
Dioptres
  Visit 1 | 0.70 (0.55) | 0.80 (0.49)
  Visit 2 | 0.45 (0.39) | 0.61 (0.33)
  Visit 3 | 0.41 (0.21) | 0.60 (0.31)

7. Secondary Outcome: Surgically Induced Astigmatism (SIA)
Description: Surgically induced astigmatism presented in dioptres at each visit.
Time Frame: Visits 4-8
Population: Surgically Induced Astigmatism-FAS Population
Measure: Mean (Standard Deviation); unit: Dioptres
Units Other Than Participants: eyes
Arm/Group | Coaxial Micro-Incision Cataract Surgery | Coaxial Small-Incision Cataract Surgery
Number analyzed (Participants) | 35 | 35
Number analyzed (eyes) | 35 | 35
Dioptres
  Visit 4 | 0.44 (0.37) | 0.52 (0.31)
  Visit 5 | 0.39 (0.36) | 0.53 (0.35)
  Visit 6 | 0.37 (0.27) | 0.59 (0.30)
  Visit 7 | 0.37 (0.31) | 0.51 (0.31)
  Visit 8 | 0.37 (0.21) | 0.42 (0.26)

ADVERSE EVENTS:
Time Frame: 12 Weeks
Description: Safety Set
Groups:
- Co-Axial Micro-Incision Cataract Surgery: 1.8 mm coaxial micro-incision cataract surgery (C-MICS) with phacoemulsification using the Stellaris Vision Enhancement System.
- Cataract Surgery All Participants: Events by participant one eye with 1.8 mm coaxial micro-incision cataract surgery (C-MICS) and the contralateral eye with the 2.75 mm coaxial standard cataract surgery.
Arm/Group | Co-Axial Micro-Incision Cataract Surgery | Coaxial Small-Incision Cataract Surgery | Cataract Surgery All Participants
Serious Adverse Events (participants affected / at risk) | 1/36 | 0/35 | 5/36
Other Adverse Events (participants affected / at risk) | 33/36 | 33/35 | 66/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-Axial Micro-Incision Cataract Surgery (N=36) | Coaxial Small-Incision Cataract Surgery (N=35) | Cataract Surgery All Participants (N=36)
Macular Degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — Pre-existing condition
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study, crossed both arms, non ocular SAE
High Blood Pressure (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study, crossed both arms, non ocular SAE
Hip Arthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study, crossed both arms, non ocular SAE
Carpal Tunnel Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study, crossed both arms, non ocular SAE
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study, crossed both arms, non ocular SAE
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-Axial Micro-Incision Cataract Surgery (N=36) | Coaxial Small-Incision Cataract Surgery (N=35) | Cataract Surgery All Participants (N=71)
Anterior Chamber Cell (Eye disorders) | 28 (30) | 30 (32) | 58 (62)
Corneal Edema (Eye disorders) | 21 (21) | 22 (22) | 43 (43)
Anterior Chamber flare (Eye disorders) | 8 (8) | 8 (9) | 16 (17)
Visual Disturbance (Eye disorders) | 4 (4) | 2 (2) | 6 (6)
Posterior Capsule Opacification (Eye disorders) | 2 (2) | 2 (2) | 4 (4)
Conjunctivitis (Eye disorders) | 2 (2) | 1 (1) | 3 (3)
Blurred Vision (Eye disorders) | 2 (2) | 1 (1) | 3 (3)
Vitreous Detachment (Eye disorders) | 2 (2) | 0 (0) | 2 (2)
Increased Intraocular Pressure (Eye disorders) | 5 (5) | 4 (4) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study data generated as a result of this study will be regarded as confidential, until appropriate analysis and review by the Sponsor or its designee and the Investigator(s) are completed. The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.